CLINICAL TRIAL: NCT03288844
Title: Multinational, Multicenter, Prospective, Long-term Safety and Efficacy Follow-up Study After Autologous Cultivated Limbal Stem Cells Transplantation (ACLSCT) for Restoration of Corneal Epithelium in Patients With Limbal Stem Cell Deficiency Due to Ocular Burns
Brief Title: Follow-up Study After ACLSCT for Restoration of Corneal Epithelium in Patients With LSCD Due to Ocular Burns
Acronym: HOLOCORE-FU
Status: Completed | Type: Observational
Sponsor: Holostem s.r.l. (Industry)
Collaborators: Cromsource (Industry)
Responsible Party: Sponsor
Other Study IDs: CCD-GPLSCD01-03-FU; 2015-001344-11 (EudraCT Number)
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Limbal Stem Cell Deficiency Due to Ocular Burn
Keywords: LSCD, Holoclar, follow-up

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HOLOCORE Patients: Patients who completed the main HOLOCORE clinical trial will undergo to Ophthalmologic examinations, Digital pictures collection and QoL questionnaires (NEI VFQ 25 and EQ-5D-3L/Y) will be performed/administered at each study visit
  Interventions: Procedure: Ophthalmologic examinations; Other: Digital pictures; Other: QoL Questionnaires

INTERVENTIONS:
Procedure: Ophthalmologic examinations — epithelial defects assessment by fluorescein staining; superficial corneal neo-vascularization assessment; ocular tonometry; slit lamp examination; conjunctival (both bulbar and limbal) inflammation assessment; corneal sensitivity; central cornea involvement (for opacity or central CNV); Best-Corrected Visual Acuity; evaluation of symptoms.
Other: Digital pictures — Digital pictures 2D to be taken at each visit
Other: QoL Questionnaires — Quality of Life (NEI VFQ 25 and EQ-5D-3L/Y) questionnaires will be submitted at each visit

SUMMARY:
This is a multinational, multicentre, prospective, non-pharmacological follow-up study of the clinical trial HOLOCORE. All patients transplanted with Holoclar in the HOLOCORE clinical trial who consent to participate will be enrolled in this prospective study and observed for at least 12 months.

DETAILED DESCRIPTION:
HOLOCORE FOLLOW-UP prospective study offers the opportunity to collect long-term efficacy and safety data after one or two treatments with Holoclar. Moreover, since Holoclar (study drug used in the main HOLOCORE interventional clinical trial) is suspected to improve the success of keratoplasty in those patients candidate to receive this treatment but no data were collected in the three previous retrospective studies (HLSTM01, HLSTM02 and HLSTM04) on Holoclar, this follow-up study has been thought to observe the progress of the disease and to collect data on keratoplasty and evaluate the benefits of Holoclar in subsequent keratoplasty in patients treated once or two times with Holoclar.

All patients treated in the HOLOCORE clinical trial who consent to roll over to the present extension study at the end of the HOLOCORE will be observed for a follow-up period which may vary from a minimum of 12 month for the last patient to a maximum of 57 months for the first patient entered.

A total of approximately 70 patients is expected (all patients who completed the HOLOCORE study).

In case the last enrolled patient undergoes to Keratoplasty at the Last Visit of the Follow-up study, this will consequently lead to a prolongation of the study up to further 12 months for all patients.

The subjects will be enrolled and observed at the same investigational centers where they were recruited for the HOLOCORE clinical trial.

No drug will be administered for the scope of this study. Ophtalmological visits including pictures collection and quality of life evaluations will be performed every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* All patients (adults and pediatrics) who completed the HOLOCORE core study and who consent to roll over to the present extension study at the end of the HOLOCORE follow-up.

Exclusion Criteria:

* No specific exclusion criterion is considered for this study, except for patients dropping out from the HOLOCORE study or withdrawing consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All eligible patients who entered the core HOLOCORE study will be asked consent to roll over into this extension study before their inclusion. Approximately 70 patients will be enrolled in this study.
  Safety population: all patients entering the study. The adult safety population will be used to explore efficacy. Efficacy data collected on paediatric population will be only listed.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Success of transplantation | 1 year
  Transplantation will be considered with a clinically-relevant success if the severity of superficial corneal neo-vascularization will be judged as not exceeding one quadrant of invasion (without central cornea involvement) by the investigator and the degree of Epithelial defect as 'None' or 'Trace', respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Graziella Pellegrini, Professor, Study Director — Holostem s.r.l.; Paolo Rama, MD, Study Chair — Fondazione I.R.C.C.S. Policlinico San Matteo, Pavia, Italy
Locations (1):
- Hospital San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No